CLINICAL TRIAL: NCT03291197
Title: Assessing the Tolerability of Suprascapular and Median Nerve Blocks for the Treatment of Shoulder-hand Syndrome - a Feasibility Study
Brief Title: Tolerability of Suprascapular and Median Nerve Blocks for the Treatment of Shoulder-hand Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20170066-01H
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Results first posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-07

CONDITIONS: Shoulder Hand Syndrome; Complex Regional Pain Syndromes
Keywords: Suprascapular nerve block; Median nerve block; CRPS; Shoulder hand syndrome
MeSH Terms: conditions — Reflex Sympathetic Dystrophy; Complex Regional Pain Syndromes | interventions — Bupivacaine; Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: Open label preliminary study testing the tolerability of the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open label treatment (Experimental): These patients will receive suprascapular and median nerve blocks for shoulder hand syndrome. Investigators will assess the tolerability of his procedure using pre-defined criteria (outlined elsewhere).
  Interventions: Drug: Suprascapular and median nerve blocks

INTERVENTIONS:
Drug: Suprascapular and median nerve blocks — Ultrasound guided injection of the median and suprascapular nerve of the affected side.
  Other Names: Bupivacaine, kenalog

SUMMARY:
Shoulder-hand syndrome (SHS) in stroke patients is painful and lowers quality of life. Unfortunately, the cause of SHS is not known, diagnosing SHS can be difficult, and treating it can be hard. Recent research has shown that certain nerve blocks are good for treating shoulder pain for stroke patients, but no one has looked specifically as SHS. Investigators think that specific nerve blocks involving a shoulder nerve (the suprascapular, or SSc nerve) and a hand nerve (the median nerve) will be helpful in reducing SHS pain. Investigators will use ultrasound guidance to accurately inject these nerves. These injections have never been described for SHS patients however, so investigators want to make sure people with SHS can go through with the injections without too much pain or discomfort. That is, the investigators want to test the tolerance of these injections for people with SHS. Investigators are also hoping to better understand how consistent a set of diagnostic criteria, called the Budapest criteria, are at diagnosing SHS in order to be able to accurately diagnose this condition.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are required to be 18 years of age or older and have a presumptive diagnosis of SHS post-stroke with a minimum visual analog scale of 40mm (greater than 40mm is considered moderate pain).

Exclusion Criteria:

* Subjects will be excluded from the study if they have significant cognitive impairment (mini-mental state examination <23) and language deficits (difficulty cooperating due to aphasia) as this may affect their response to the outcome measures. Subjects with uncontrolled hypertension (>180/110), septicemia, and brachial plexus injuries will be excluded. Patients who are blind and deaf will also be excluded, as they will be unable to adequately complete the post-procedure survey and VAS. Patients on anticoagulation medications will also be excluded on a case-by-case basis and medications will be held prior to injection if required for safety. Patients with INR >1.5 will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2018-10-14 (Actual); Study Completion 2018-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: T Mark Campbell, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Elisabeth Bruyere Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was from September 2017 to 2018. This was a 12 month period in which patient with shoulder and hand pain following stroke were recruited.
Pre-assignment Details: All participants were recruited to for suprascapular and median nerve blocks once a diagnosis of shoulder-hand-syndrome was made using the Budapest criteria
Groups:
- Open Label Treatment: These patients received suprascapular and median nerve blocks for shoulder hand syndrome. Investigators assessed the tolerability of his procedure using pre-defined criteria (outlined elsewhere).
  Suprascapular and median nerve blocks: Ultrasound guided injection of the median and suprascapular nerve of the affected side.
Period: Overall Study
Arm/Group | Open Label Treatment
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Open Label Treatment: These patients will receive suprascapular and median nerve blocks for shoulder hand syndrome. Investigators will assess the tolerability of his procedure using pre-defined criteria (outlined elsewhere).
  Suprascapular and median nerve blocks: Ultrasound guided injection of the median and suprascapular nerve of the affected side.
  Outcome measure were recorded for each participant before, immediately after, and 2 weeks post intervention.
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 5
Right Hand Dominant [Count of Participants; unit: Participants] | 5
Mini Mental Status Exam [Mean (Standard Deviation); unit: units on a scale] — Cognitive test. Total score out of 30 points. A total score below 24 is considered cognitively impaired. We are not including subscales and report only on the total score.
  units on a scale | 26.6 (1.1)
Stroke Location [Count of Participants; unit: Participants]
  Right middle cerebral artery | 2
  Right posterior limb of internal capsule | 2
  Left pons | 1
Time interval, days [Mean (Standard Deviation); unit: Days] — The number of days from the date of study enrolment to the date the participants received peripheral nerve injections.
  Days | 12.8 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Demonstrating Tolerability of Suprascapular and Median Nerve Blocks
Description: To evaluate the tolerability of ultrasound-guided suprascapular and median nerve blocks in stroke patients with SHS as determined using the Budapest criteria. Since tolerability is a subjective measure, it will be defined by a composite outcome including: A) Pain score prior to, during, and immediately following the procedure as measured by the visual analog scale (VAS); B) the rate of serious adverse events associated with this procedure; and C) the level of patient acceptance and satisfaction as determined by a validated post-procedure survey.
Time Frame: 12 months
Population: All participants tolerated the intervention
Measure: Count of Participants; unit: Participants
Groups:
- Tolerability: Composite score of: a) change in VAS by > 18mm; b) rate of serious adverse events; c) level of patient satisfaction
Arm/Group | Tolerability
Number analyzed (Participants) | 5
Participants | 5

2. Primary Outcome: Visual Analog Scale (VAS)
Description: Pain scale used to address a difference following intervention. Pain is measured on a horizontal line from 0 to 100mm, with 0 being no pain and 100 being the worst imaginable pain. Participants place a vertical mark on the line indicating their pain intensity.
Time Frame: measured at baseline, within 1 hour after, and 2 weeks post intervention
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Baseline VAS: visual analog pain scale at baseline prior to intervention
- 1 Hour VAS: VAS measured within 1 hour after intervetion
- 2 Weeks VAS: VAS measured 2 weeks post intervention
Arm/Group | Baseline VAS | 1 Hour VAS | 2 Weeks VAS
Number analyzed (Participants) | 5 | 5 | 5
score on a scale
  Shoulder | 75 [66.5 to 90.5] | 17 [0 to 29.5] | 22 [0 to 63]
  Hand | 36 [24.5 to 80.5] | 16 [0 to 32.5] | 28 [0 to 57]
Statistical Analysis 1: Comparison: Baseline VAS vs 1 Hour VAS; Our study was not powered to perform statistical analysis though was still conduct to look for a trend in reduction of VAS; Test type: Other; p = 0.043, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Inter-rater Agreement of Budapest Criteria
Description: Investigators will assess the reproducibility of the Budapest clinical criteria for newly suspected cases of SHS. This will be achieved by determining the level of inter-rater agreement between a resident and a staff physician working in stroke rehabilitation. Investigators will thus determine if there is variability in the clinical diagnosis among physicians with different levels of expertise.
Time Frame: 12 months
Measure: Number; unit: Intraclass correlation coefficient
Groups:
- All Participants: All participants will be assessed using the Budapest Criteria by both a staff physician and a resident. The inter-rater agreement will be determined to assess the reproducibility of the Budapest clinical criteria for newly suspected cases of SHS.
Arm/Group | All Participants
Number analyzed (Participants) | 5
Intraclass correlation coefficient | 0.75

ADVERSE EVENTS:
Time Frame: during and immediately following the procedure
Groups:
- Tolerability: Composite score
Arm/Group | Tolerability
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
Some of these results should be considered hypothesis-generating due to the small sample size of our study, and the inability to assess other factors that may affect the response to pain (i.e. co-morbidities, psychological profile).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT03291197/Prot_SAP_000.pdf